CLINICAL TRIAL: NCT02246465
Title: An Open-Label, Multi-Center, Prospective, Within-Subject Controlled, Phase 2a Study to Evaluate the Effectiveness and Safety of RXI 109 on the Outcome of Scar Revision Surgery for Hypertrophic Scars in Healthy Adults
Brief Title: A Study to Evaluate the Effectiveness and Safety of RXI 109 on the Outcome of Revised Hypertrophic Scars
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RXi Pharmaceuticals, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXI-109-1402
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Hypertrophic Scar
Keywords: Hypertrophic scar; Cicatrix; Scar prevention; Scar revision
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RXI-109 (Experimental): RXI-109 dosed at the site of the revised hypertrophic scar
  Interventions: Drug: RXI-109

INTERVENTIONS:
Drug: RXI-109

SUMMARY:
The purpose of this study is to determine the effectiveness of RXI-109 in reducing the recurrence of hypertrophic scar formation following elective revision of a pre-existing hypertrophic scar.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21-55 years of age
* General good health
* Previous surgery or injury resulting in a hypertrophic scar

Exclusion Criteria:

* Scars on the face or front of neck may not be included in the trial
* Use of tobacco or nicotine-containing products
* Pregnant or lactating

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Reducing the recurrence of hypertrophic scar after scar revision surgery | 9 months
  To evaluate the effectiveness of RXI-109 in reducing the recurrence of hypertrophic scar formation following elective scar revision surgery by review of photographic results and Patient and Observer Scar Assessment Scales.

SECONDARY OUTCOMES:
Safety evaluation of RXI-109 | 9 months
  To assess severity and frequency of reported adverse events and clinically-relevant changes in laboratory testing after elective revision of a hypertrophic scar

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Pavco, PhD, Study Director — RXi Pharmaceuticals
Locations (6):
- United States (5):
  - Beverly Hills, California
  - Lake Worth, Florida
  - Chicago, Illinois
  - St Louis, Missouri
  - Huntersville, North Carolina
- San Pedro Sula, Honduras